CLINICAL TRIAL: NCT04279691
Title: Synovial and Gingival Crevicular Fluid Levels of Prolactin Hormone in Rheumatoid Arthritis Patients With Periodontitis
Brief Title: Prolactin Hormone in Rheumatoid Arthritis Patients With Periodontitis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: October University for Modern Sciences and Arts (Other)
Responsible Party: Principal Investigator, Naglaa Elwakeel, professor, October University for Modern Sciences and Arts
Other Study IDs: ETH14
Record Dates: First submitted 2020-02-19; First posted 2020-02-21 (Actual); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: Rheumatoid Arthritis; Periodontitis
MeSH Terms: conditions — Arthritis, Rheumatoid; Periodontitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Synovial fluid and gingival crevicular fluid
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- periodontitis and rheumatoid arthritis: group 1: patiernts with periodontitis and rheumatoid arthritis. only
- periodontitis: group 2: patiernts with periodontitis

SUMMARY:
In this study we will assess the presence of prolactin hormone in the gingival crevicular fluid , and synovial fluid of patient with rheumatoid arthritis and periodontitis

ELIGIBILITY:
Inclusion Criteria:

* for first group patients with active rheumatoid arthritis with periodontitis.
* second group , patients with periodontitis and otherwise systemically healthy
* third group, systemically and periodontallly healthy subjects

Exclusion Criteria:

* smokers,
* pregnant or lactating females
* patients taking medications the affects levels of prolactin hormone.
* no periodontal treatment in the past six months

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Egyptian patients with active rheumatoid arthritis and periodontitis.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-03 (Estimated); Primary Completion 2020-04 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
prolactin hormone levels in the tested media | 24 hours
  changes in prolactin hormone expression in the tested media

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] El-Wakeel NM, Shalaby ZF, Abdulmaguid RF, Elhamed SSA, Shaker O. Local gingival crevicular fluid, synovial fluid, and circulating levels of prolactin hormone in patients with moderately active rheumatoid arthritis and stage III and IV periodontitis before and after non-surgical periodontal treatment-a controlled trial. Clin Oral Investig. 2023 Jun;27(6):2813-2821. doi: 10.1007/s00784-023-04867-w. Epub 2023 Jan 31. PMID 36717425